CLINICAL TRIAL: NCT07274553
Title: The Effect of a Mindfulness-Based Stress Reduction Program on Digital Game Addiction Levels, Perceived Stress, and Sleep Quality in Adolescents
Brief Title: Mindfulness-Based Stress Reduction for Adolescents: Effects on Game Addiction, Stress, and Sleep
Acronym: MBSR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/461
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Adolescent Behaviour Disorder; Stress Reduction; Sleep Quality; Digital Addiction
Keywords: Mindfulness-Based Stress Reduction; Adolescents; Digital Game Addiction; Nursing; Stress; Sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to an intervention group that received an 8-week Mindfulness-Based Stress Reduction (MBSR) program and a control group that received no intervention. The study followed a two-arm, parallel-group, pretest-posttest design.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Mindfulness-Based Stress Reduction (MBSR) (Experimental): Participants in this group will receive an 8-week Mindfulness-Based Stress Reduction (MBSR) program specifically designed for adolescents. Each session lasts approximately 40 minutes and includes breathing awareness, body scan, mindful movement, and emotional regulation exercises. The sessions are conducted once a week in a classroom setting by a trained instructor. Participants are encouraged to practice mindfulness exercises at home between sessions.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction Program (MBSR)
- No Intervention: Control Group (No Intervention): Participants in this group will not receive any mindfulness or behavioral intervention. They will continue their normal school routine and educational activities during the study period. After the study concludes, they will be offered a brief introductory mindfulness session as an ethical consideration.

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction Program (MBSR) — The intervention consists of an 8-week Mindfulness-Based Stress Reduction (MBSR) program adapted for adolescents. Each weekly session lasts approximately 40 minutes and is conducted in a classroom setting by a trained instructor. The program includes breathing awareness, body scan, mindful movement, and emotion regulation exercises. Participants are encouraged to practice mindfulness at home between sessions using simple guided exercises.
  Arms: Experimental: Mindfulness-Based Stress Reduction (MBSR)

SUMMARY:
This randomized controlled trial investigated the impact of a Mindfulness-Based Stress Reduction (MBSR) program on digital game addiction, perceived stress, and sleep quality among adolescents. The primary research questions were as follows: Does the Mindfulness-Based Stress Reduction Program influence adolescents' levels of digital game addiction? Does the Mindfulness-Based Stress Reduction Program affect adolescents' perceived stress levels? Does the Mindfulness-Based Stress Reduction Program impact adolescents' sleep quality? Participants, aged 12-16, will be randomly allocated to either an intervention group, which will undergo an 8-week MBSR program, or a control group, which will continue with routine school activities. The MBSR program comprises weekly 40-minute sessions that include breath awareness, body scanning, mindful movement, and emotion regulation exercises. Data will be collected using the Digital Game Addiction Scale, Perceived Stress Scale, and Pittsburgh Sleep Quality Index at both the pretest and posttest stages. This study is anticipated to contribute to the development of preventive strategies for behavioral addictions and enhance the emotional well-being and sleep patterns of adolescents.

DETAILED DESCRIPTION:
The Mindfulness-Based Stress Reduction (MBSR) program is a structured behavioral intervention aimed at enhancing awareness and emotional regulation through mindfulness practices. This study assessed the efficacy of an 8-week MBSR program implemented in high school settings in Muş, Turkey. A total of 80 adolescents (40 intervention and 40 control) will voluntarily participate in the study. The intervention group will engage in mindfulness sessions concentrating on "being present," "breath awareness," "accepting difficult emotions," and "self-compassion." Each session will have a duration of approximately 40 min per week. Ethical approval was obtained from the Atatürk University Non-Interventional Clinical Research Ethics Committee (Decision No: 2025/461). The anticipated findings aim to provide evidence supporting the use of mindfulness-based interventions to enhance adolescent mental health and prevent digital gaming addiction.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged between 12 and 16 years
* Enrolled in a high school under the Muş Provincial Directorate of National Education
* Voluntarily agreed to participate and provided informed consent (along with parental consent)
* Able to attend all eight weeks of the mindfulness sessions
* Sufficient literacy and comprehension to complete self-report questionnaires

Exclusion Criteria:

* Diagnosed psychiatric, neurological, or developmental disorder
* Currently receiving psychological therapy or participating in another behavioral program
* Regular use of medication that affects sleep, mood, or cognitive function
* Absence from more than two MBSR sessions
* Declined or withdrew consent during the study period

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2025-11-03 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Digital Game Addiction Score | Baseline (Week 0) and Post-intervention (Week 8)
  Measured by the Digital Game Addiction Scale. Score range: 7 (minimum) to 35 (maximum). Higher scores indicate worse outcomes, representing higher levels of digital game addiction.

SECONDARY OUTCOMES:
Perceived Stress Score | Baseline (Week 0) and Post-intervention (Week 8)
  Measured by the Perceived Stress Scale. Score range: 0 (minimum) to 56 (maximum). Higher scores indicate worse outcomes, reflecting a higher level of perceived stress.
Sleep Quality Score | Baseline (Week 0) and Post-intervention (Week 8)
  Measured by the Pittsburgh Sleep Quality Index. Score range: 0 (minimum) to 21 (maximum). Higher scores indicate worse outcomes, representing poorer sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University, Health Sciences Institute, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No